CLINICAL TRIAL: NCT06972602
Title: High-dose Topotecan for Retinoblastoma With Recurrent or Refractory Vitreous Seed(A Prospective Non-controlled Single Arm Trial)
Brief Title: High-dose Topotecan for Retinoblastoma With Recurrent or Refractory Vitreous Seed
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-EENT-2018044-1
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Retinoblastoma; Retinoblastoma, Recurrent
MeSH Terms: conditions — Retinoblastoma; Recurrence | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-dose Topotecan for Retinoblastoma With Recurrent or Refractory Vitreous Seed (Experimental): Intravitreal injection of topotecan at a dosage of 100μg was performed on day 1 of week 1.The frequency of treatment is personalized by ophthalmologists based on the intraocular stage of RB and treatment response. The criteria for end event are complete disappearance of vitreous seeding or stable calcification. Patients were followed up and evaluated every four weeks, with collection of aqueous humor and electroretinogram examination.
  Interventions: Drug: Topotecan; Other: Collection of aqueous humor; Other: Electroretinogram

INTERVENTIONS:
Drug: Topotecan — Intravitreal injection of topotecan at a dosage of 100μg was performed at week 1.Then based on the tumor response and vitreous seeding, it will be decided whether to continue the injection by ophthalmologists.
Other: Collection of aqueous humor — Patients' aqueous humor samples will be collected for Inflammatory factor testing and IOP control every 4 weeks.
Other: Electroretinogram — Electroretinogram was performed every 4 weeks.

SUMMARY:
Retinoblastoma is the most common intraocular malignancy in infancy and childhood,with an estimated 8000 new cases globally each year.The major cause of failure in the management of retinoblastoma remains the persistence or recurrence of resistant vitreous seeding.Currently,with the emergence of new administration routes, intravitreal chemotherapy has been used for vitreous seeds and the rate of eye preservation has been effectively improved. However, the use of high doses of chemotherapeutic agents may lead to visual impairments due to long term retinal toxicity and some tumors recur or become resistant to chemotherapeutic agents after treatment. In such cases, ocular resection is the only option to prevent extraocular metastasis and death.

Therefore, studies on retinoblastoma are currently focused on finding new targeted therapies at appropriate doses to increase anti-tumor activity and reduce side effects. In this study, Topotecan at a dosage of 100μg will be used to treat patients with refractory or recurrent retinoblastoma.

On one hand, topotecan, as a topoisomerase I inhibitor, prevents the reconnection of broken single stranded DNA, causing irreversible DNA damage. On the other hand, topotecan upregulates PTEN protein to restore its inhibitory effect on the PI3K/AKT signaling pathway, thereby jointly promoting tumor cell apoptosis and weakening cell proliferation activity.Topotecan at a dosage of 100μg has been proven safe in animal experiments, and there have been a few retrospective case reports on its application in retinoblastoma, but relevant prospective clinical studies are still lacking.

Based on the above background, this study will explore the feasibility and effectiveness of intravitreal injection of Topotecan at a dosage of 100μg in patients with refractory or recurrent retinoblastoma through a prospective study,while evaluating immune response and visual preservation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with retinoblastoma with a somatic mutation of the gene RB1 and active tumor in a single eye, or germinal mutation of RB1 with active tumor/s in an eye and the contralateral eye unaffected, enucleated or without tumor activity. In both cases, relapsed or refractory vitreous seeding with the use of systemic, intraarterial or intravitreal chemotherapy or radiotherapy, in accordance with the availability at his/her referral site, in whom enucleation is the only recommended treatment under opinion of the medical team treating the case at the originating referral site. But the patient has a strong desire to preserve the eye.
2. Normal renal function: serum creatinine: < 45 μmol/L (0-2 years); < 57 μmol/L (3-6 years); < 60 μmol/L (7-10 years); < 80 μmol/L (11-13 years).
3. Normal Hepatic function: serum ALT: < 0,52 μkat/L (de 9 months -12 years); serum AST: 61-80 g/L (8 months-5 years); 63-83 g/L (5-9 years); 63-82 g/L (9-12 years).
4. Adequate marrow reserve manifested in an absolute neutrophil count > 1000 / mm3, platelets > 100,000 / mm3 and hemoglobin> 8 g / dl, without transfusional or cytokine support at least one month prior to study entry.
5. Age greater than 1 year and less than 12 years at the time of inclusion in the study.
6. Sign the informed consent form and be willing to follow up at the specified time.

Exclusion Criteria:

1. Presence of factors that require immediate enucleation of the affected eye such as glaucoma, rubeosis iridis, anterior chamber involvement.
2. Comorbidities: Uncontrolled epilepsy with anticonvulsant treatment, cardiac disease not compensated by treatment.
3. Active Infections.
4. Other chronic or active acute diseases that under the criterion of the researcher were an exclusion criterion.
5. History of having received attenuated or live vaccines in the 30 days prior to inclusion in the study.
6. Any cause of Immunosuppression.
7. Trilateral Retinoblastoma.
8. Extraocular spread.
9. History of having received treatment for retinoblastoma with chemotherapy or radiation therapy by any means within 30 days prior to inclusion in the study.
10. Patients who can not complete the study procedures for reasons psychologically or socially

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 28 days
  Tumor response rate (ORR) to Topotecan at 28 days post-administration.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 13 weeks
Immune response | 13 weeks
  Inflammatory factor testing was performed on the patients' aqueous humor samples.
Electroretinogram | 13 weeks
  Electroretinogram was performed to evaluate patient's retinal function and visual preservation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Eye & ENT Hospital, Shanghai, China, China